CLINICAL TRIAL: NCT05968027
Title: Improving Care Pathway Using Simplified Digital Tools for Oncology Patients: a Multicenter "Before-and-after" Study
Acronym: ONCONECTSAFE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Nouveal (Unknown)
Responsible Party: Sponsor
Other Study IDs: APHP230641
Record Dates: First submitted 2023-07-21; First posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Oncology; Adverse Event; Numeric Application; Care Telemonitoring; Compliance, Treatment; Patient Reported Outcome (PRO)
MeSH Terms: conditions — Neoplasms; Patient Compliance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Onco'nect pre-deployment: - Onco'nect pre-deployment (12 months): period covering the year prior to the actual implementation of the solution in each centre; patients receiving I.V. chemotherapy during the first 6 months of the period will be included, in order to assess the 6-month follow-up.
- Onco'nect post-deployment: -Onco'nect post-deployment (12 months): period covering the year following the implementation of the solution within the centre (installation, interoperability and parameterisation validated); patients with I.V. chemotherapy implemented during the first 6 months of the period will be included, in order to be able to evaluate the 6-month follow-up.
  Interventions: Other: Nouveal numeric application "Onco'nect"

INTERVENTIONS:
Other: Nouveal numeric application "Onco'nect" — A remote monitoring application, Onco'nect® (smartphone /tablet /PC), in partnership with the company Nouveal facilitates communication between patients undergoing Intra Vascular (IV) chemotherapy and the care team. A questionnaire before and after each session can be used to alert the oncology department and adapt patient management.
  Groups: Onco'nect post-deployment

SUMMARY:
Developments in the healthcare sector in general, and in oncology in particular, mean that patients are increasingly autonomous. Outpatient treatment raises the issue of home monitoring. One of the solutions proposed by the 2014-2019 Cancer Plan is the development of telemedicine. Several programmes have been set up in the medical oncology department at Hôpital Mondor, to make patient care more secure and improve the management of undesirable effects of treatment for patients undergoing intravenous (I.V.) chemotherapy or oral anti-cancer treatments.

The preliminary study on the use of the digital solution Onco'nect demonstrated the feasibility of using a dematerialised tool for real-time monitoring and management of chemotherapy-induced adverse events in cancer patients undergoing outpatient treatment. The tool was used to help AP-HP institution deal with the crisis linked to the COVID epidemic. Once it had been configured, Onco'nect was deployed to all institution's hospital groups to ensure that infected patients could remain at home, and that patients hospitalised with symptomatic COVID infection could return home.

Hypothesis: The digital solution Onco'nect would improve patient compliance and could reduce the occurrence and improve the management of unexpected adverse events.

Primary objective:

In terms of clinical evaluation, the primary objective is to assess the effect of using the Onco'nect solution for ambulatory oncology follow-up on reducing the rate of occurrence at 6 months follow-up of unexpected and unwanted chemo-induced adverse events.

The solution is already on the market and has been integrated (or is in the process of being integrated) into the care systems of the participating AP-HP establishments. The aim of the project is to evaluate its use in routine care and measure the occurrence and management of unexpected and unwanted chemo-induced adverse events in outpatients treated for cancer.

This observational study of care pathway, using retrospective data, aims to include 480 patients in a 18 months period.

Three periods of interest will be considered in this before-and-after study

* Onco'nect pre-deployment (12 months): period covering the year prior to the actual implementation of the solution in each centre; patients receiving I.V. chemotherapy during the first 6 months of the period will be included, in order to assess follow-up at 6 months.
* Onco'nect deployment: this period corresponds to the implementation of the solution in the centre's care pathway. Deployment includes interoperability with other operating systems and setting up the collection interfaces for the user.
* Post-deployment (12 months): period covering the year following the implementation of the solution within the centre (installation, interoperability and configuration validated); patients receiving I.V. chemotherapy during the first 6 months of the period will be included, in order to be able to evaluate the 6-month follow-up.

ELIGIBILITY:
Inclusion criteria

* Age >=18 years
* Initiation of I.V. chemotherapy for solid cancer of any location or metastatic status:
* Either over a period of 12 months before Onco'nect is deployed, covering the year preceding the actual implementation of the solution in each centre.
* Or over a period of 12 months post-deployment of Onco'nect, covering the year following the implementation of the solution within the centre.
* Non-opposition to the study and to the processing of their medical data.

Exclusion criteria

* Any known difficulty in understanding or reading French that might invalidate the relevance of applying questionnaires
* Known cognitive or psychiatric disorder preventing the protocol from being carried out
* Patient under legal protection
* Patient included in the article 51 programme

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients treated with IV chemotherapy and monitored in the medical oncology departments of participating centres (AP-HP): CHU Henri Mondor Créteil (HMN), CHU Pitié Salpêtrière Paris (PSL), CHU Bichat Paris (BCT), CHU Saint Antoine (SAT) and CHU Georges Pompidou (HEGP).
Sampling Method: Probability Sample
Enrollment: 480 (Estimated)
Dates: Start 2024-01-02 (Estimated); Primary Completion 2025-07-02 (Estimated); Study Completion 2025-07-02 (Estimated)

PRIMARY OUTCOMES:
adverse events | during a 6 months follow-up period starting after chemotherapy injection
  presence of one or more unexpected and undesirable chemo-induced adverse events at 6 months' follow-up after the start of chemotherapy (use of unscheduled hospitalisation, consultation/admission to the emergency department, grade 3 and 4 toxicities according to version 5 of the CTCAE, changes in chemotherapy administration schedules, such as last-minute cancellations, changes in dose and frequency of treatment administration).

CONTACTS AND LOCATIONS:
Overall Officials: Christophe TOURNIGAND, MD-PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris

IPD SHARING:
Plan to Share IPD: No
AP-HP, as sponsor, is the owner of the data and no use or transmission to a third party may be made without its prior agreement.